CLINICAL TRIAL: NCT06250478
Title: Het Gebruik Van Dynamische Echografie om Spier-pees Veranderingen te Onderzoeken in de Kuitspieren Van Personen na Een CVA: Een Pilootstudie
Brief Title: Dynamic Ultrasound of the Calf Muscles After Stroke
Acronym: Stroke_DynUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2023-0497; B6702023000632 (Registry Identifier: Belgium register)
Record Dates: First submitted 2024-01-17; First posted 2024-02-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Gait Disorders, Neurologic
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Both stroke patients and age and gender matched healthy controls will be included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patient (Experimental)
  Interventions: Diagnostic Test: Dynamic ultrasound of the calf muscles
- Healthy controls (Active Comparator)
  Interventions: Diagnostic Test: Dynamic ultrasound of the calf muscles

INTERVENTIONS:
Diagnostic Test: Dynamic ultrasound of the calf muscles — Dynamic changes of the calf muscles during walking will be assessed in persons after stroke and compared to healthy controls

SUMMARY:
Muscle behaviour of calf muscles can be studied during dynamic conditions using dynamic ultrasound. In particular, the medial gastrocnemius is suitable for measurements with dynamic ultrasound due to its superficial location. With this measurement technique, the muscle behavior during walking can be observed gaining insight into the mechanism of action of this muscle during a functional task. This technique has already been used in other populations (such as children with cerebral palsy) but not yet in individuals after a stroke.

Therefore, the aim of this study is to assess the muscle behavior of the medial gastrocnemius during walking in persons after stroke. There are 3 concrete objectives of the current study:

1. is the technique feasible to perform in persons after stroke?
2. does the use of the dynamic echoprobe change gait patterns?
3. can differences between persons after stroke and healthy controls be detected? This data can be used as pilot data for project applications in the future that will allow to design larger studies.

Therefore, 10 stroke patients and 10 age- and gender-matched healthy controls will walk on a treadmill for 3x2 minutes after a familiarisation period of 6 minutes.

During 1 x 2 minutes, subjects will walk without using the dynamic ultrasound. This recording aims to measure the normal gait pattern of the subjects.

During the other 2x2 minutes, subjects will walk using the dynamic ultrasound at 2 different locations on the calf. Once with the ultrasound probe on the centre of the muscle belly to visualise muscle fibre bundles and once on the muscle tendon transition, from which muscle belly and tendon length can be derived.

The use of ultrasound or not will be randomized to exclude the effect of fatigue on the outcome measures.

ELIGIBILITY:
Stroke group Inclusion criteria

* stroke adults
* no other neurologic conditions
* ability to walk independently on a treadmill

Exclusion criteria

* wearing ankle foot orthosis that inhibit the assessment
* had lower limb surgery in the past

Healthy volunteers Inclusion criteria

- healthy adults

Exclusion criteria

* suffering from any neurological condition
* had lower limb surgery in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Fascicle dynamics measured with ultrasound during walking | single point assessment in one day during walking with the probe
  Lengthening and shortening of the fascicles of the medial gastrocnemius
Muscle belly dynamics measured with ultrasound during walking | single point assessment in one day during walking with the probe
  Lengthening and shortening of the muscle belly of the medial gastrocnemius
Tendon dynamics measured with ultrasound during walking | single point assessment in one day during walking with the probe
  Lengthening and shortening of the tendon of the medial gastrocnemius

SECONDARY OUTCOMES:
gait speed | single point assessment in one day during walking with the probe
  walking velocity (m/s)
gait speed | single point assessment in one day during walking without the probe
  walking velocity (m/s)
step width | single point assessment in one day during walking with the probe
  step width (m)
step width | single point assessment in one day during walking without the probe
  step width (m)
Step length | single point assessment in one day during walking with the probe
  Step length (m) of the paretic and non paretic side
Step length | single point assessment in one day during walking without the probe
  Step length (m) of the paretic and non paretic side
stance phase | single point assessment in one day during walking with the probe
  time spend standing on the paretic and non-paretic leg (s) during walking
stance phase | single point assessment in one day during walking without the probe
  time spend standing on the paretic and non-paretic leg (s) during walking
swing phase | single point assessment in one day during walking with the probe
  time spend not standing on the paretic and non-paretic leg (s) during walking
swing phase | single point assessment in one day during walking without the probe
  time spend not standing on the paretic and non-paretic leg (s) during walking
lower limb kinematics | single point assessment in one day during walking with the probe
  joint angles (°) in the pelvis, hip, knee and ankle in the sagittal, frontal and transverse plane during walking
lower limb kinematics | single point assessment in one day during walking without the probe
  joint angles (°) in the pelvis, hip, knee and ankle in the sagittal, frontal and transverse plane during walking

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No